CLINICAL TRIAL: NCT01883739
Title: Randomised Controlled Trial to Investigate the Effect of Parental Presence at Intensive Care Unit to Ward Transfer Bedside Rounds on Parental Anxiety and Children's Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Medical Protective Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro 00037475
Record Dates: First submitted 2013-06-17; First posted 2013-06-21 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Parental Anxiety; Children's Safety
Keywords: Parental anxiety; Children's safety; Family Centered Care; Bedside Transfer Rounds; Pediatric Cardiac Intensive Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parental Presence at Handover Rounds (Experimental): Subjects will receive an educational document prior to transfer rounds introducing the concept of Patient and Family Centered Care and the role of a parent in transfer rounds. These parents will have the option of meeting with a parental peer support person for a "coaching" or training session prior to their participation in transfer rounds. During the transfer rounds parents will be actively included in discussion of their child's medical management plan upon discharge to the wards.
  Interventions: Other: Parental Presence at Handover Rounds

INTERVENTIONS:
Other: Parental Presence at Handover Rounds

SUMMARY:
The investigators shall conduct a randomized controlled trial to investigate the effect of parental presence at transfer rounds on parental anxiety and patient safety following transfer from the Pediatric Cardiac Intensive Care Unit (PCICU) to the ward. The investigators plan to test the hypothesis that parental involvement in the child's transfer, with the option of peer support, will result in measurable reductions in medication errors, unplanned nutritional and feeding management, and parental anxiety after transfer as compared to the control group. The investigators goal is to improve continuity of care by implementing multidisciplinary transfer rounds at the child's bedside in which patients and family share in the control of the management plan when a cardiac child is discharged from PCICU to the ward.

ELIGIBILITY:
Inclusion Criteria:

* Parents of cardiac children aged 1 day to 17 years admitted to PCICU
* Written informed consent and assent when appropriate
* Planned discharge from the PCICU to the ward.

Exclusion Criteria:

* Parents with less than grade 6 reading skills as they will not be able to independently take the Spielberger's State -Trait Anxiety Inventory (STAI).
* Parents who are not willing to be randomized to the control group in which they cannot be present for transfer rounds.
* Neonates being discharged from PCICU to NICU or neonates being discharged from NICU to wards.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in parental STAI score | 2 to 4 hours post transfer
  Speilberger State-Trait Anxiety Inventory will be administered to participating parents both prior to and post transfer of their child out of the pediatric cardiac ICU.

SECONDARY OUTCOMES:
Rate of unplanned changes in medication and nutrition management | 48 hours post transfer
  Medication and nutritional order reconciliation will occur 48 hours after transfer from the PCICU. The pharmacist, dietician and physician who review the patient charts and order sheets will be blinded to the randomization. Differences between pre and post transfer orders will be discussed to detect omissions and/or deviation from standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Adatia, MBChB, MRCP, FRCP(C), Principal Investigator — Stollery Children's Hospital, University of Alberta
Locations (1):
- Pediatric Cardiac ICU, Stollery Children's Hospital, Edmonton, Alberta, Canada